CLINICAL TRIAL: NCT01796574
Title: Feasibility and Tolerability of the Ketogenic Diet in the Treatment of Refractory Status Epilepticus in a Neurointensive Care Unit.
Brief Title: Ketogenic Diet for Refractory Status Epilepticus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Mayo Clinic (Other); Queen's Medical Center (Other); Rush University Medical Center (Other); Oregon Health and Science University (Other); Thomas Jefferson University (Other); Intermountain Medical Center (Other); NYU Langone Health (Other); University of Rochester (Other)
Responsible Party: Principal Investigator, Mackenzie Cervenka, Assistant Professor of Neurology, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00073063
Record Dates: First submitted 2013-01-11; First posted 2013-02-22 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Status Epilepticus; Seizure; Epilepsy; Refractory Status Epilepticus; Medically Resistant Status Epilepticus
Keywords: status epilepticus; seizure; epilepsy; ketogenic diet; modified Atkins diet
MeSH Terms: conditions — Status Epilepticus; Seizures; Epilepsy | interventions — Diet, Ketogenic; Fluid Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ketogenic diet (Experimental): Patients will receive the ketogenic diet as a formula delivered via feeding tube. Once able to tolerate food by mouth, patients will be switched to a modified Atkins diet.
  Interventions: Dietary Supplement: Ketogenic diet

INTERVENTIONS:
Dietary Supplement: Ketogenic diet — 4:1 ratio fat: carbohydrates and protein ketogenic liquid via enteral feed
  Other Names: KetoCal 4:1 liquid

SUMMARY:
This research is being done to observe the safety, tolerability, side effects, and effectiveness of the ketogenic diet in people with continuous seizures (status epilepticus) being treated in a neurointensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older in refractory status epilepticus (continuous or recurrent seizures without return to baseline mental status between seizures, lasting > 30 minutes) placed on anesthetics/sedating agents (barbiturates or benzodiazepines) after at least one first- and second-line agent failed to control seizures, and with clinical and/or electrographic seizures following attempt to wean anesthetic/sedating agents after 24 hours.

Exclusion Criteria:

1. Unstable metabolic condition
2. Hemodynamic or cardiorespiratory instability
3. Coagulopathy
4. Liver failure
5. Total cholesterol > 300 mg/dL
6. Inability to tolerate enteral feeds, including ileus
7. Pregnancy
8. Family refusal/no consent
9. Received any propofol infusions within 24 hours
10. Known fatty acid oxidation disorder or pyruvate carboxylase deficiency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-11; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Feasibility | 2 weeks
  Whether or not the diet protocol was followed

SECONDARY OUTCOMES:
Time to seizure reduction | Participants will be followed for the duration of the hospital stay, an expected average of 6 weeks
  The time (in days) from initiation of the diet to > 50% reduction in frequency and to resolution of electrographic (based on continuous EEG findings) and/or clinical seizures will be recorded.
Ranking of tolerability measures on a 10 point scale | 6 months
  Participants will complete a scale ranking convenience, taste, texture, tolerance
Number of participants with adverse events and description of events | 6 months
  Reported side effects will be recorded as well as number of patients who develop side effects.
Time to achieving serum and/or urinary ketosis | Until serum or urinary ketosis is achieved, an expected average of 2 weeks
  The time (in days) from starting the ketogenic diet to achieving urinary and/or serum ketosis will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Mackenzie C. Cervenka, MD, Principal Investigator — Johns Hopkins University
Locations (9):
- United States (9):
  - Mayo Clinic, Phoenix, Arizona
  - Queen's Medical Center, Honolulu, Hawaii
  - Rush University Medical Center, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - New York University, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Intermountain Medical Center, Murray, Utah

REFERENCES:
- [Background] Vaccarezza M, Silva W, Maxit C, Agosta G. [Super-refractory status epilepticus: treatment with ketogenic diet in pediatrics]. Rev Neurol. 2012 Jul 1;55(1):20-5. Spanish. PMID 22718405
- [Background] Ferlisi M, Shorvon S. The outcome of therapies in refractory and super-refractory convulsive status epilepticus and recommendations for therapy. Brain. 2012 Aug;135(Pt 8):2314-28. doi: 10.1093/brain/aws091. Epub 2012 May 9. PMID 22577217
- [Background] Nam SH, Lee BL, Lee CG, Yu HJ, Joo EY, Lee J, Lee M. The role of ketogenic diet in the treatment of refractory status epilepticus. Epilepsia. 2011 Nov;52(11):e181-4. doi: 10.1111/j.1528-1167.2011.03289.x. Epub 2011 Oct 17. PMID 22003821
- [Background] Nabbout R, Mazzuca M, Hubert P, Peudennier S, Allaire C, Flurin V, Aberastury M, Silva W, Dulac O. Efficacy of ketogenic diet in severe refractory status epilepticus initiating fever induced refractory epileptic encephalopathy in school age children (FIRES). Epilepsia. 2010 Oct;51(10):2033-7. doi: 10.1111/j.1528-1167.2010.02703.x. Epub 2010 Aug 31. PMID 20813015
- [Background] Cervenka MC, Hartman AL, Venkatesan A, Geocadin RG, Kossoff EH. The ketogenic diet for medically and surgically refractory status epilepticus in the neurocritical care unit. Neurocrit Care. 2011 Dec;15(3):519-24. doi: 10.1007/s12028-011-9546-3. PMID 21523523
- [Background] Wusthoff CJ, Kranick SM, Morley JF, Christina Bergqvist AG. The ketogenic diet in treatment of two adults with prolonged nonconvulsive status epilepticus. Epilepsia. 2010 Jun;51(6):1083-5. doi: 10.1111/j.1528-1167.2009.02388.x. Epub 2009 Oct 20. PMID 19845731
- [Background] Thakur KT, Probasco JC, Hocker SE, Roehl K, Henry B, Kossoff EH, Kaplan PW, Geocadin RG, Hartman AL, Venkatesan A, Cervenka MC. Ketogenic diet for adults in super-refractory status epilepticus. Neurology. 2014 Feb 25;82(8):665-70. doi: 10.1212/WNL.0000000000000151. Epub 2014 Jan 22. PMID 24453083
- See also: Adult Epilepsy Diet Center at Hopkins website — http://www.hopkinsmedicine.org/neurology_neurosurgery/specialty_areas/epilepsy/adult/adult-epilepsy-diet-center/